CLINICAL TRIAL: NCT07263373
Title: Multicenter Cohort Study on Predicting Bronchiectasis Progression, Complications, and Prognosis Through Multimodal Integration of Radiomics, Clinical Features, and Lung Microbiota
Brief Title: Multicenter Cohort Study on Predicting Bronchiectasis Progression, Complications, and Prognosis Using Multi-omics
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-SR-695
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Bronchiectasis Adult; Radiomics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bronchiectasis

SUMMARY:
Bronchiectasis is a heterogeneous condition with diverse etiologies and clinical manifestations. Its progression involves a vicious cycle of airway inflammation, recurrent infection, and structural damage, leading to persistent symptoms and declining lung function. Current management focuses on airway clearance and antibiotics, with no disease-modifying therapies available. Recognizing this heterogeneity is crucial for advancing targeted treatments and precision medicine.

Radiomics converts medical images into mineable data to reveal underlying pathophysiology. While applied in other respiratory diseases, its potential in bronchiectasis remains underexplored. Both radiomics and the lung microbiome are independently linked to disease severity in conditions like COPD, but their interplay is unclear. Integrating these modalities with clinical data could unlock novel insights, identify new therapeutic targets, and improve diagnostic and prognostic models.

However, few studies have investigated multimodal models combining radiomics, microbiome, and clinical features to predict outcomes in bronchiectasis. To address this gap, we designed a multicenter, retrospective study. It will analyze data from patients diagnosed between January 2020 and July 2025 to evaluate the combined value of radiomics, microbial features, and clinical parameters in diagnosing and predicting the progression of bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* ① Diagnosis of bronchiectasis;

  * Availability of both raw high-resolution computed tomography (HRCT) chest images and the corresponding radiology report; ③ Age ≥ 18 years.

Exclusion Criteria:

* ① Incomplete clinical data;

  * Absence of chest CT imaging studies and reports; ③ Other patients deemed ineligible for enrollment at the investigator's discretion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of bronchiectasis established by high-resolution CT (HRCT) of the chest and its corresponding radiology report.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
death | 2025.7

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University，, Nanjing, Jiangsu, China